CLINICAL TRIAL: NCT07192068
Title: Widening Treatment Options Among Adult Patients With HER2-overexpressing or Mutant Solid Cancers.
Brief Title: Clinical Trial Evaluating the Activity of Zanidatamab for the Treatment of Patients With Solid Tumors With an Alteration of the HER2 Gene.
Acronym: AcSé HER2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: National Cancer Institute, France (Other Government); Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-GMP-2505; 2025-522169-31-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-21; First posted 2025-09-25 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer; Sarcoma; Head &Amp; Neck Cancer; Colorectal Carcinoma; Endometrial
Keywords: zanidatamab; HER2 mutant; HER2-IHC3+
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Sarcoma; Head and Neck Neoplasms; Colorectal Neoplasms | interventions — zanidatamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- zanidatamab (Experimental): Single arm study where the experimental regimen used for all patients will be zanidatamab, administered intravenously every 3 weeks :
  * Patients <70 kg: 1800 mg IV Q3W on Day 1 of each 21-day cycle
  * Patients ≥70 kg: 2400 mg IV Q3W on Day 1 of each 21-day cycle.
  Interventions: Drug: Zanidatamab

INTERVENTIONS:
Drug: Zanidatamab — Single arm study where the experimental regimen used for all patients will be zanidatamab, administered intravenously every 3 weeks :
  * Patients <70 kg: 1800 mg IV Q3W on Day 1 of each 21-day cycle
  * Patients ≥70 kg: 2400 mg IV Q3W on Day 1 of each 21-day cycle.

SUMMARY:
Alterations in the HER2 gene are involved in the development of cancer. These abnormalities are found at highly variable rates (from approximately 2% to 60%) in cancers of the lung, breast, stomach, bile ducts, salivary glands, colon, endometrium, uterus, bladder, bones, blood, etc. Zanidatamab is an anti-cancer drug that acts on cells with alterations in the HER2 gene. It is used in Europe to treat people with bile duct cancer.

However, in various clinical trials, zanidatamab has shown promising activity in a few patients with different cancers that have a HER2 gene alteration. This treatment could therefore be effective in several types of cancer once this gene alteration is detected.

The primary objective is to evaluate the efficacy of zanidatamab in patients with cancer in one of the following locations: endometrium, colorectal, head and neck, sarcoma or lung cancer. Efficacy will be measured by the number of patients in whom a reduction in tumour size was observed.

All patients included in the study will receive zanidatamab by intravenous infusion every 3 weeks. Treatment will continue as long as there is a benefit (stabilisation or regression of the disease). During treatment, participants will visit the hospital regularly for medical consultations to:

* assess and treat potential adverse effects of zanidatamab. A dose reduction may be applied to improve tolerance.
* monitor disease progression using scans and/or MRI, performed every 6 weeks for the first 18 months of treatment and then every 12 weeks.

After treatment is stopped (due to intolerance or disease progression), patients will be monitored according to hospital practices until the end of the trial, i.e. for 1 to 4 years, depending on when they were included in the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed endometrial, colorectal, head & neck, non-small cell lung cancer (NSCLC), or sarcoma
2. Patient with progressive, unresectable and/or advanced or metastatic disease harboring a locally performed, centrally reviewed HER2-overexpressing (IHC 3+ exclusively) for endometrial, colorectal, head & neck cancers, or sarcoma or a HER2 activating mutation for NSCLC, determined on tissue (see Section 7.1.2 of the protocol)
3. Age ≥ 18 years at inclusion
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
5. Patient who progressed at least after 1 line of therapy, for whom there is no other standard therapeutic option available
6. Patient with a HER2 alteration covered by a standard marketed indication for any HER2 targeting therapy should be included after standard anti-HER2 strategy has been exhausted.
7. Estimated life expectancy >3 months
8. Measurable disease according to RECIST1.1, whatever the disease location. Tumor lesions located in a previously irradiated area, or in an area subjected to other loco-regional therapy, are considered measurable if progression has been clearly demonstrated in the lesion
9. Adequate bone marrow function: absolute neutrophil count (ANC) ≥1.5 × 10⁹/L, platelet count ≥75 × 10⁹/L, and haemoglobin ≥9 g/dL. Transfusion is allowed with a 2-week washout period before treatment initiation
10. Adequate liver function: total bilirubin level ≤1.5 × the upper limit of normal (ULN) range (total bilirubin ≤3.0 ULN when the patient has documented Gilbert syndrome or liver metastasis), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤2.5 × ULN (AST and ALT ≤5 ULN when documented tumor liver involvement)
11. Adequate cardiac function: left ventricular ejection fraction (LVEF) ≥ 50% at baseline as determined by either echocardiogram (ECHO) or multigated acquisition (MUGA) scan within 14 days before inclusion
12. Normal prothrombin time (PT) >70% and partial thromboplastin time (PTT), except for patient who uses anticoagulants
13. Adequate renal function: estimated serum creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula
14. Man, and woman of childbearing potential must agree to use highly effective contraception for the duration of trial participation and as required after completing study treatment (refer to Table 6 in the protocol). Man must also agree to not donate sperm and women must agree to not donate oocytes during the specified period
15. Woman of childbearing potential must have a negative serum pregnancy test performed within 3 days before the date of treatment initiation
16. Availability of a suitable archived FFPE sample of primary or metastatic tumor tissue (archived FFPE is <2 years old (desirable), maximum 5 years (accepted), buffered formalin fixed only. Fine-needle aspiration (cytology samples) and biopsies from sites of bone metastases are not acceptable) or patient accepts an optional biopsy under study
17. Willing and able to comply with the protocol for the duration of the study including scheduled visits, treatment plan, laboratory tests, specimen sampling for research, and other study procedures
18. Affiliated to a social security system
19. Patient must have signed a written informed consent form prior to any trial specific procedures. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in signing the patient's consent.

Exclusion Criteria:

1. Patient, in the judgment of the investigator, who should be included in another recruiting study assessing an anti-HER2 therapy (including zanidatamab)
2. Patient who received prior treatment with HER2-directed therapy unless marketed for the study cohort indication.
3. Other primary malignancies within 3 years with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin. Cancer survivor, who has undergone potentially curative therapy for a prior malignancy, has no evidence of that disease for 4 years or more and is deemed at negligible risk for recurrence, is eligible for the trial
4. Any autoimmune, connective tissue or inflammatory disorder with pulmonary involvement not related to lung metastases (e.g. rheumatoid arthritis, Sjögren's syndrome, sarcoidosis)
5. Prior pneumonectomy
6. Patient with any condition or any evidence of severe or uncontrolled systemic diseases (e.g. active bleeding diatheses, active infection, or psychiatric illness) which in the investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardize compliance with the protocol. Screening for chronic conditions is not required for eligibility
7. History of myocardial infarction or unstable angina within 6 months prior to enrolment, troponin levels consistent with myocardial infarction, or clinically significant cardiac disease, such as ventricular arrhythmia requiring therapy, uncontrolled hypertension, or any history of symptomatic congestive heart failure
8. Evidence of spinal cord compression or brain metastases, defined as being clinically active and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Patient with clinically inactive or treated brain metastases who are asymptomatic (i.e. without neurologic signs or symptoms and do not require treatment with corticosteroids or anticonvulsants) may be included in the study. Patient must have a stable neurologic status and no evidence of radiographic progression for at least 2 weeks prior to first zanidatamab dosing
9. Patient with evidence of any leptomeningeal disease. If leptomeningeal disease has been reported radiographically on baseline magnetic resonance imaging (MRI), but is not suspected clinically by the investigator, the subject must be free of neurological symptoms.
10. Acute or chronic uncontrolled pancreatitis or Child-Pugh Class C liver disease
11. Patient with unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to grade ≤1 or baseline, as defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Patient with chronic Grade 2 toxicities may be enrolled at the discretion of the investigator after consultation and approval by the coordinating investigator.
12. Patient receiving chronic systemic corticosteroids dosed at >10 mg prednisone or equivalent anti-inflammatory activity or any form of immunosuppressive therapy within 2 weeks of first zanidatamab dosing unless otherwise approved by the coordinating investigator. Patient who requires use of bronchodilators, inhaled or topical or ocular steroids, or local steroid injections may be included in the study
13. Treatment with anthracyclines within 90 days before first dose of zanidatamab and/or total lifetime load exceeding 360 mg/m2 doxorubicin or equivalent
14. A history of life-threatening hypersensitivity to monoclonal antibodies or recombinant proteins
15. Woman who is pregnant or breast-feeding
16. Participation in another therapeutic trial within the 30 days prior to entering the study. Participation in an observational trial would be acceptable
17. Patient unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons
18. Individual deprived of liberty or placed under protective custody or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2028-03-13 (Estimated); Study Completion 2030-06-24 (Estimated)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate (ORR) by investigator | From Baseline to disease progression (up to 28 months)
  Confirmed Objective Response Rate (ORR) for each cohort, based on best overall response, defined as the percentage of patients with a complete response (CR) or partial response (PR) during treatment or follow-up, assessed according to RECIST1.1, by investigator assessment and confirmed by a follow-up scan at ≥ 4 weeks from first response assessment.

SECONDARY OUTCOMES:
Confirmed ORR by the BICR | From baseline to the progression (up to 28 months)
  Confirmed ORR for each cohort, based on best overall response as adjudicated by the BICR, defined as the percentage of patients with a CR or PR during treatment or follow-up, assessed according to RECIST1.1 and confirmed by a follow-up scan at ≥ 4 weeks from first response assessment
Duration of Response (DoR) | From baseline to the progression (up to 28 months)
  Duration of Response (DoR) for each cohort will be evaluated in patients with either a CR or PR. DoR is defined as the time from the first assessment of a confirmed CR or PR until the date of the first occurrence of progressive disease (PD) according to RECIST1.1 or death from any cause (if death occurs within predefined period), whichever occurs first. At the time of analysis, a patient alive and without disease progression will be censored at the date of the last valid tumor assessment. DoR will be provided as assessed by investigators and as adjudicated by the BICR.
Progression Free Survival (PFS) | From baseline to disease progression or death (up to 28 months)
  Progression Free Survival (PFS) for each cohort is defined as the time from study registration until disease progression (per RECIST1.1) or death from any cause, whichever occurs first. At the time of analysis, a patient alive and without disease progression will be censored at the date of the last valid tumor assessment. PFS will be provided as assessed by investigators and as adjudicated by the BICR.
Clinical Benefit Rate (CBR) | From baseline to the progression (up to 28 months)
  Clinical Benefit Rate (CBR) for each cohort is defined as the percentage of patients with a CR or PR or stable disease (SD) for more than 16 weeks from inclusion assessed according to RECIST1.1. CBR will be provided as assessed by investigators and as adjudicated by the BICR.
Overall Survival (OS) | From baseline to death (up to 52 months)
  Overall Survival (OS) for each cohort is defined as the time from study registration until death from any cause. Patients who are alive at last follow-up will be censored at this date.
Incidence of treatment-Emergent Adverse Events [Safety and Tolerability of zanidatamab] | From baseline to the end of treatment (up to 28 months)
  The safety will be evaluated according to the incidence of adverse events (AEs) graded by NCI-CTCAE v5.0, per cohort and overall.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara PISTILLI, Dr, Principal Investigator — Gustave Roussy, VILLEJUIF
Locations (4):
- France (4):
  - Institut de Cancérologie de l'Ouest, Angers
  - Chu Timone, Marseille
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.